CLINICAL TRIAL: NCT00536458
Title: Phase III Study of Treatment of Localized Lymphomas: Radiotherapy Versus Radio-Chemotherapie
Brief Title: Treatment of Localized Low Grade Lymphomas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01 02; GOELAMS 01 02; GOELNH LOGLOC
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-09

CONDITIONS: Lymphoma, Low-Grade
Keywords: localized low grade lymphoma; Chemotherapy; Radiotherapy; Molecular analyses; primary
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- radiotherapy (Experimental): minichep + radiotherapy
  Interventions: Procedure: radiotherapy
- B (Active Comparator): MINI CHEP
  Interventions: Drug: MINI CHEP

INTERVENTIONS:
Procedure: radiotherapy — mini chep+ radiotherapy
  Arms: radiotherapy
Drug: MINI CHEP — chemotherapy minichep 6 courses
  Arms: B

SUMMARY:
To compare localiezd radiotherapy to localized radiotherapy followed by 6 cycles of chemotherapy in the treatment of localiezd low grade lymphoma

DETAILED DESCRIPTION:
The standard treatment ol localized low grade lymphomas is Radiotherapy alone can offer long term remissions to some patients .

No study have clearly demonstrated the interest of chemotherapy. The purpose of the study is to determine wether prednisone administrated after first line local radiotherapy (30 GY) can pre in the treatment of localized low grade lymphomas of adult patients

ELIGIBILITY:
Inclusion Criteria:

* Low grade lymphoma defined according to the Ann Arbor classification
* localized

Exclusion Criteria:

* Subjects unable to signed informed consent
* Pregnancy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 1999-03; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
failure free survival at 5 years | 5 years

SECONDARY OUTCOMES:
overall survival at 5 years | 5 years
response rates at the end of the treatment | 6 months
prognstic value of molecular analyses in blood and marrow | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: eric DECONINCK, MD PhD, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- Regional university hospital, Besançon, France